CLINICAL TRIAL: NCT04839640
Title: Study of Wear in Composite Resin and Reinforced Acrylic Denture Teeth Used in Complete Denture Construction for Completely Edentulous Patients (Randomized Controlled Trial)
Brief Title: Study of Wear in Composite Resin and Reinforced Acrylic Denture Teeth Used in Complete Denture Construction for Completely Edentulous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shereen ismail, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 123456789
Record Dates: First submitted 2018-04-17; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Wear, Occlusal
MeSH Terms: conditions — Tooth Attrition

STUDY DESIGN:
Intervention Model Description: split mouth technique
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reinforced acrylic resin denture teeth (Active Comparator): Shufo acrylic denture teeth
  Interventions: Other: Bredent denture teeth
- Composite resin denture teeth (Experimental): Bredent denture teeth
  Interventions: Other: Bredent denture teeth

INTERVENTIONS:
Other: Bredent denture teeth — composite resin denture teeth

SUMMARY:
Visit 1: Clinical examination and investigations will be carried out for the eligible patients including TMJ examination and intraoral examination for oral mucosa. Diagnostic charts will be prepared with full medical and dental history as well as radiographic records. Primary impression will be performed with irreversible hydro-colloid impression material (alginate), The impressions will be poured with type IV dental stone to obtain diagnostic casts, special tray will be constructed.

Visit 2: Maxillary Face-bow will be recorded to mount the upper cast. The diagnostic casts will be mounted on semi adjustable articulator in centric occluding relation to evaluate the inter-arch distance.

Visit 3: Secondary impression will be performed in special trays by elastomeric impression material. The impression will be poured into typeIV dental stone in order to obtain master cast.

Visit 4: Trial denture base will be constructed and tried in patient's mouth for obtaining maxilla-mandibular relation using face bow record and centric relation record, then mounting of the casts on semi adjustable articulator will be done. The teeth will be set according to the randomization group.

Visit 5: The denture bases will be tried in with acrylic teeth in patient's mouth.

Visit 6: The denture will be delivered to the patient and occlusal adjustments will be done.

Visit 7: Recall visit after one week, further adjustments will be done. The denture will be sent to the scanning center and given to the patient again.

Visit 8: At 3 months follow up, the denture will be inspected for calculus and will be immersed in ultrasonic cleaner for 15 seconds to remove calculus and then scanned.

Visit 9: At 6 months follow up, the denture will be inspected for calculus and will be immersed in ultrasonic cleaner for 15 seconds to remove calculus and then scanned.

Visit 10: At 9 months follow up, the denture will be inspected for calculus and will be immersed in ultrasonic cleaner for 15 seconds to remove calculus and then scanned.

The optical methods tend to fulfill the need for quantitative characterization of surface topography. Specimens will be photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X.The images will be recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images will be cropped using Microsoft office picture manager to specify/standardize area of roughness measurement. The cropped images will be analyzed using WSxM software. Specimens will be photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X. The images will be recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images will be cropped to 350 x 400 pixels using Microsoft office picture manager to specify/standardize area of roughness measurement. The cropped images will be analyzed using WSxM software.

ELIGIBILITY:
Inclusion Criteria:

Edentulous subjects with indication for full dentures Skeletal class I maxillomandibular relationship

Exclusion Criteria:

Uncooperative patients. Subjects that wear dentures for less than 6 hours per day Subjects from which no compliance can be expected

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Optical scanning to detect difference in wear at baseline and 3 months follow up visits | 3 months
  Specimens will be photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X. The images will be recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images will be cropped to 350 x 400 pixels using Microsoft office picture manager to specify/standardize area of roughness measurement. The cropped images will be analyzed using WSxM software.
Optical scanning to detect difference in wear at baseline and 6 months follow up visits | 6 months
  Specimens will be photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X. The images will be recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images will be cropped to 350 x 400 pixels using Microsoft office picture manager to specify/standardize area of roughness measurement. The cropped images will be analyzed using WSxM software.
Optical scanning to detect difference in wear at baseline and 9 months follow up visits | 9 months
  Specimens will be photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X. The images will be recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images will be cropped to 350 x 400 pixels using Microsoft office picture manager to specify/standardize area of roughness measurement. The cropped images will be analyzed using WSxM software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided